CLINICAL TRIAL: NCT03477747
Title: Efficacy of Microcurrent to Maximise Exercise Outcomes, Accelerate Recovery and Attenuate Muscle Damage in Athletes
Brief Title: The Application of Microcurrent in Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Greenwich (Other)
Collaborators: Arc Family (Unknown)
Responsible Party: Principal Investigator, Fernando Naclerio, Associate Professor, University of Greenwich
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UREC/16.3.5.13
Record Dates: First submitted 2018-03-18; First posted 2018-03-26 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Training Group, Sensitivity
Keywords: Microcurrent; Exercise training; Hypertrophy; Muscle damage; Recovery; Performance
MeSH Terms: conditions — Hypersensitivity; Hypertrophy

STUDY DESIGN:
Intervention Model Description: Double-blind randomise controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind (Subject, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Resistance Training Microcurrent (Experimental): Participants will combine a 10-week periodized and controlled resistance programme with 3 h of microcurrent after training.
  Measurements pre and post-intervention will be body composition via DEXA, endurance performance (1 RM bench press and Squat) endurance (vo2max) and blood markers: haemoglobin; red blood cell; erythrocyte; haematocrit; mean corpuscular volume, transferrin; neutrophils; lymphocyte; monocytes, IL6, IL1, Myoglobin, salivary cortisol and testosterone. Elbow flexors, vastus medialis and vbastus lateralis muscle thickness
  Interventions: Device: Microcurrent
- Resistance Training Shadow (Sham Comparator): Participants will combine a 10-week periodized and controlled resistance programme with 3 h of sham comparator after training.
  Measurements pre and post-intervention will be body composition via DEXA, endurance performance (1 RM bench press and Squat) endurance (vo2max) and blood markers: haemoglobin; red blood cell; erythrocyte; haematocrit; mean corpuscular volume, transferrin; neutrophils; lymphocyte; monocytes, IL6, IL1, Myoglobin, salivary cortisol and testosterone. Elbow flexors, vastus medialis and vbastus lateralis muscle thickness
  Interventions: Device: Microcurrent
- Endurance Training Microcurrent (Experimental): Participants will combine a 10-week periodized and controlled endurance programme with 3 h of microcurrent after training.
  Measurements pre and post-intervention will be body composition via DEXA, endurance performance (1 RM bench press and Squat) endurance (vo2max) and blood markers: haemoglobin; red blood cell; erythrocyte; haematocrit; mean corpuscular volume, transferrin; neutrophils; lymphocyte; monocytes, IL6, IL1, Myoglobin, salivary cortisol and testosterone. Elbow flexors, vastus medialis and vbastus lateralis muscle thickness
  Interventions: Device: Microcurrent
- Endurance Training Shadow (Sham Comparator): Participants will combine a 10-week periodized and controlled endurance programme with 3 h of microcurrent after training.
  Measurements pre and post-intervention will be body composition via DEXA, endurance performance (1 RM bench press and Squat) endurance (vo2max) and blood markers: haemoglobin; red blood cell; erythrocyte; haematocrit; mean corpuscular volume, transferrin; neutrophils; lymphocyte; monocytes, IL6, IL1, Myoglobin, salivary cortisol and testosterone. Elbow flexors, vastus medialis and vbastus lateralis muscle thickness
  Interventions: Device: Microcurrent

INTERVENTIONS:
Device: Microcurrent — Microcurrent based treatments have been proposed more than 30 years. The manufacturer initially should calibrate the microcurrent devices. There is no physical sensation associated with microcurrent based treatments as the strength of the current is not high enough to stimulate sensory nerve fibres. The application of electric fields and currents similar to those generated within the body can substantially change the cell structure and the metabolic behaviour of cells. For example, the application of microcurrent increases the number of organelles responsible for cellular activities; it increases concentrations of adenosine triphosphate (ATP) and amino acid transport; promotes protein synthesis; fastens regrowth of atrophied soleus muscle and would also activate hormone-sensitive lipase which can increase lipolysis from the internal and external adipose tissue. The microcurrent treatment with training would maximize exercise and recovery outcomes in athletes.

SUMMARY:
The aim of this investigation is to analyse the potential benefits of wearing a new commercially available microcurrent device combined with different exercise training modalities on exercise outcomes, body composition, recovery including muscle damage, general markers of health and immune function in athletes.

DETAILED DESCRIPTION:
The investigation involves two randomised, balanced, double-blind parallel group between-participants design, aimed to analyse the effects of combining microcurrent with resistance and endurance training. Participants, once considered eligible for the study will be familiarised with the respective exercises, as well as tested for baseline values. Thereafter participants will be randomly assigned to one of the following intervention groups (1) Microcurrent (MCR+RT) with resistance training (2) Microcurrent (MCR+END) with endurance training (3) Sham with resistance training (SH+RT) and (4) Sham with endurance training (SH+END). Participants will perform 3 supervised training sessions per week (24 total workouts). Participants will wear the microcurrent or sham devices during 3 hr after workouts. Each group will follow a 10-week resistance or endurance training intervention combined with one of the two specific treatments (MCR or SH). Measurements of body composition, muscle thickness, performance, salivary and blood markers as well as delayed onset of muscle soreness will be determined before and after each particular (resistance or endurance training) intervention.

Participants It is anticipated that sixty participants, recruited from the Medway University Campus, will take part in the project. Inclusion criteria are: regularly trained male or female athletes, aged 18 to 45 years old, with at least 3 months of experience in resistance or endurance training, with no musculoskeletal injuries, metabolic conditions, or diseases or use of medications, smoking, and nutritional supplements known to affect physical performance, muscle damage or recovery processes (e.g., creatine, whey protein, and amino acids, vitamin or mineral supplementation, etc) within 6 weeks prior to the start of the study.

After being informed of all risks and potential benefits involved, participants will sign a written informed participation consent form. Procedures will be in accordance with the Helsinki Declaration and will be approved by the Research Ethics Committee of the University of Greenwich.

Intervention Resistance training groups

Familiarization period:

Participants will undertake 3 sessions of familiarization (1 week). To ensure a correct execution of the selected exercise a qualified strength and conditioning coach will control and assists participants. All participants will be instructed about the appropriate use of the Rate of Perceived Exertion OMNI-RES (0-10) scale to control the load and training intensity during each workout.

The resistance-training program is designed to increase strength and muscle mass of all major muscle groups. Under the supervision of strength and conditioning coaches, preferable a MSc Strength and Conditioning student from the University of Greenwich. The program will be undertaken on three non-consecutive days per week, Training workout will be performed during the afternoon (between 3 pm and 6 pm) with at least 48 hours between sessions.

The intervention period consists of a 8-week periodised resistance training programme divided into 3 blocks: First block (week 1 to week 3) using a moderate load intensity of around 70% 1RM; Second block (week 4 to week 6) where the intensity increases to >75% to 80% 1RM and the third block (week 7 to week 8) where the highest loads (>80 to 85% 1RM) are implemented. The Rate of Perceive Exertion OMNI-RES (0-10) scale (RPE) will be used to appropriately select the loading zone for each particular exercise during the workouts (Naclerio et al., 2015a, Naclerio et al., 2011)

Each workout session begins with individualized warm-up (5-minute warm-up stretches, followed by one set of eight repetitions of six resistance training exercises without any additional weight). Workouts will involve 3 sets of 8 to 10 RM (self maximal estimation) with approximately 2 min of rest of the following exercises:

1. Parallel back squat
2. Hang clean
3. Alternate lunges with dumbbells
4. Bench press
5. Upright row
6. Double leg dead lift
7. Push Press
8. Front shoulder press and
9. Biceps curl.

Each workout will last between 45 to 60 min.

The load will be increased or decrease based on the self-perception of the participants. When a minimum of 8 Reps is no possible to complete the participants will rest for 15sec and complete the set. Additionally, the participants can decide to reduce the load for the next set. Conversely, when more than 10 reps can be performed, the participants will stop the set, increase the load and complete the 10RM set.

Endurance training Participants will commit to follow a polarised triphasic endurance-training model. This model contains three intensity zones calculated as low intensity [≥ the first ventilatory threshold (VT1), ~ 70% HRmax]; moderate intensity [between VT1 and respiratory compensation point or ventilatory threshold 2 (VT2), >70 < 90% HRmax]; and high intensity [>VT2, 90% HRmax] (Esteve-Lanao et al., 2007). Participants will train 4 to 6 times per week with a total percentage distribution of 75 to 80% at low intensity; 10% at moderate intensity, and 15 to 10% at high intensity. Participants have to be completed the same time exposure to the MCR or SH device after the end of the intervention period.

Microcurrent or shadow

Both the microcurrent and sham devices will look exactly the same in terms of appearance, colour, size and weight. As the current transmitted from the microcurrent device is insufficient to stimulate sensory nerve fibres, this stimulus is imperceptible and together with the same appearance, participants nor strength and conditioning coaches or researchers involved in testing will be able to identify participants under the MCR or the SH treatment. Only one researcher not involved in the assessment and training supervision will know the participant allocation during the study.

Microcurrent or sham devices will be codified and placed on the participants before each training session. The participants will remove the device 10 to 15 min after completing each training session and return it to the strength and conditioning coach.

ELIGIBILITY:
Inclusion Criteria:

* Regularly trained endurance or strength athletes
* Minimum of 6 months of experience

Exclusion Criteria:

* Musculoskeletal injuries, metabolic diseases
* Use of medications
* Smoking
* Consuming any nutritional supplements that potentially affect physical performance (e.g., creatine, whey protein, and amino acids) within 6 weeks prior to the start of the study

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Body composition | 10 weeks
  Fat mass
Body composition | 10 weeks
  Fat Free Mass
Endurance Performance | 10 weeks
  Vo2 max
Strength Performance | 10 weeks
  Maximal strength
Blood Markers | 10 weeks
  haemoglobin
Blood Markers | 10 weeks
  haematocrit
Salivary markers | 10 weeks
  Cortisol
Salivary Markers | 10 weeks
  HNP1-3

SECONDARY OUTCOMES:
Hypertrophy | 10 weeks
  Muscle Thickness
Muscle Damage | 10 weeks
  Interleukin 1
Muscle Damage | 10 weeks
  Interleukin 6
Muscle Damage | 10 weeks
  Myoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Naclerio, Ph D, Principal Investigator — University of Greenwich
Locations (1):
- Department of Life and Sports Science, Eltham, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided